CLINICAL TRIAL: NCT06193096
Title: Evaluation of the Impact of a Probiotic-based Formula on Digestive Symptoms, General Symptoms and Mood in Ultra Runners
Brief Title: Impact of a Probiotic-based Formula on Digestive Symptoms and Mood in Ultra Marathon Runners
Acronym: AB-ULTRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AB Biotics, SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AB-ULTRA
Record Dates: First submitted 2023-12-21; First posted 2024-01-05 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-01

CONDITIONS: Signs and Symptoms
Keywords: Gastrointestinal symptoms; exercise; probiotics
MeSH Terms: conditions — Signs and Symptoms; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Randomized, prospective, double-blind, placebo-controlled
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Probiotic formula, 1 stick/day
  Interventions: Dietary Supplement: Experimental product
- Control group (Placebo Comparator): Placebo formula, 1 stick/day
  Interventions: Dietary Supplement: Control product

INTERVENTIONS:
Dietary Supplement: Experimental product — Probiotic mix (i3.1) comprising Pediococcus acidilactici KABPTM 021, Lactiplantibacillus plantarum KABPTM 022 and Lactiplantibacillus plantarum KABPTM 023 in a 1:1:1 ratio and with a total concentration of ≥3x10^9 total colony forming units (CFU) per sachet (stick). Other ingredients are dextrose and maltodextrin as excipients, aroma, flavorings and silicon dioxide. Experimental product will be taken over 4 weeks.
  Arms: Experimental group
Dietary Supplement: Control product — Placebo product containing dextrose and maltodextrin, aroma, flavorings and silicon dioxide.
  Control product will be taken over to weeks
  Other Names: Placebo
  Arms: Control group

SUMMARY:
Randomized, prospective, double-blind, placebo-controlled study in ultramarathon runners to evaluate the effects of suplementation with i3.1 probiotic formulation on the relief of common digestive symptoms associated to intense physical exercise. Secondary study outcomes aim to evaluate the effect of the probiotic formulation on fatigue, discomfort and muscle pain, as well as anxiety and mood.

DETAILED DESCRIPTION:
Gastrointestinal symptoms (GIS) are a common feature of intense exercise, especially in ultra-endurance events. The main objective of this study is to evaluate the impact of a 3-strain probiotic formulation comprising Lactiplantibacillus plantarum and Pediococcus acidilactici on digestive symptoms in a maximum of 300 runners registered in an organized ultra-marathon event. A randomized, prospective, double-blind, placebo-controlled study will be conducted. Once recruited, participants will be allocated to recieve either the probiotic or placebo (at a ratio 2:1) for 4 weeks prior to race day. During follow-up, study participants will fulfill several questionnaires at specific time points (baseline, week -3, -2, -1, -24 h previous to the race, as well as 24 h and 7 days after the race). This will be documented through a specifically designed, web-based platform. Digestive symptoms will be evaluated through validated questionnaires: modified from Pfeiffer et al (2012; main outcome) and the Gastrointestinal Symptoms Rating Scale (GSRS). Secondary objectives will comprise anxiety, mood, other symptoms (muscle pain, fatigue, respiratory symptoms), and performance in the ultra-marathon.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Correctly registered in the Salomon Ultra Pirineu 100K® 2023 race
* Stable medication planned during the study period
* Willing to provide informed consent and follow study procedures
* Have signed the consent provided by the organization of the Salomon Ultra Pirineu 100K® 2023 race

Exclusion Criteria:

* Respiratory, gastrointestinal or systemic infection that has caused fever or fatigue in the 15 days prior to the study entry
* Having taken probiotic-based supplements or dairy products with probiotics (including "Actimel" or yogurts with "bifidus") daily in the 15 days prior to the study start
* Taking oral or parenteral antibiotics in the 15 days prior to the study start
* History of gastrointestinal surgery within 6 months prior to the study start
* History of cardiovascular event: angina, heart failure, myocardial infarction
* Diabetes mellitus type 1 or 2
* Pregnancy or lactation, or women planning to conceive during the study period
* Chronic gastrointestinal disease: inflammatory bowel disease (Crohn's disease, ulcerative colitis), pancreatitis, short bowel syndrome
* Gastrointestinal disease or disorders: inflammatory bowel disease (ulcerative colitis, Crohn's disease), irritable bowel syndrome, chronic diarrhea or constipation
* Diagnosis of severe kidney disease (chronic kidney failure) or liver disease (hepatitis, cholestasis, liver failure)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Digestive symptoms associated to physical exercise | Baseline, +24 hours after race
  Digestive tract digestive symptoms score measured with modified Pfeiffer questionnaire. Scoring ranges from 0 to 10 according to the intensity of the symptom (0-2 non-existent or mild symptoms; 3-7 moderate symptoms; 8-10 severe symptoms)

SECONDARY OUTCOMES:
Digestive symptoms - subscore general digestive discomfort | Baseline, +24 hours after race
  Evaluation of general digestive discomfort measured with modified Pfeiffer questionnaire. Scoring ranges from 0 to 10 according to the intensity of the symptom (0-2 non-existent or mild symptoms; 3-7 moderate symptoms; 8-10 severe symptoms)
Digestive symptoms - subscore upper gastrointestinal symptoms | Baseline, +24 hours after race
  Evaluation of upper gastrointestinal symptoms subscore measured with modified Pfeiffer questionnaire. Scoring ranges from 0 to 10 according to the intensity of the symptom (0-2 non-existent or mild symptoms; 3-7 moderate symptoms; 8-10 severe symptoms)
Digestive symptoms - subscore lower gastrointestinal symptoms | Baseline, +24 hours after race
  Evaluation of lower gastrointestinal symptoms subscore measured with modified Pfeiffer questionnaire. Scoring ranges from 0 to 10 according to the intensity of the symptom (0-2 non-existent or mild symptoms; 3-7 moderate symptoms; 8-10 severe symptoms)
Digestive symptoms - subscore other gastrointestinal symptoms | Baseline, +24 hours after race
  Evaluation of other gastrointestinal symptoms (nausea, dizziness, stitch) subscore measured with modified Pfeiffer questionnaire. Scoring ranges from 0 to 10 according to the intensity of the symptom (0-2 non-existent or mild symptoms; 3-7 moderate symptoms; 8-10 severe symptoms)
Digestive symptoms - percentage of severity | Baseline, +24 hours after race
  Percentage of participants with severe symptoms (value >4) measured with modified Pfeiffer questionnaire. Scoring ranges from 0 to 10 according to the intensity of the symptom (0-2 non-existent or mild symptoms; 3-7 moderate symptoms; 8-10 severe symptoms)
Digestive symptoms measured with GSRS | week -3, -2 and -1 previous race,-24 hours before race, +7 days after race
  Evaluation of digestive symptoms measured with Gastrointestinal Symptom Rating Scale (GSRS) questionnaire. The GSRS has a 7-point graded Likert-type scale where 1 represents absence of troublesome symptoms and 7 represents very troublesome symptoms
Competitive Anxiety before race | -24 hours (before race)
  Score of the Competitive State Anxiety Inventory-2R (CSAI-2R) questionnaire. The scoring ranges from 0 (nothing) to 4 (a lot).
Race time | +24 hours after the race
  Race time at the end of the ultra in participants who finalize the race
Abandonment during the race | +24 hours after the race
  Percentage of abandonment during the race for any reason (including gastrointestinal problems)
Stool consistency | -24 hours before race, +24 hours after race
  Evaluation of stool consistency measured through Bristol scale (score from 1 to 7). Types 1 and 2 indicate constipation, with 3 and 4 being the ideal stools as they are easy to defecate while not containing excess liquid, 5 indicating lack of dietary fiber, and 6 and 7 indicate diarrhoea
Mood States | +24 hours, +7 days (after race)
  Score of the total Profile of Mood States (POMS) and the associated factors: Tension, Depression, Anger, Vigor, and Fatigue, evaluated using a visual analogue scale (VAS). The scoring ranges from 0 (not at all) to 4 (extremely).
Muscle pain | -24 hours before race, +24 hours after race, +7 days
  Muscle pain, evaluated through Visual Analogue Scale (VAS) scale. The scoring ranges from 0 (not at all) to 10 (extremely).
Fatigue | -24 hours before race, +24 hours after race, +7 days
  Fatigue, evaluated through Visual Analogue Scale (VAS) scale. The scoring ranges from 0 (not at all) to 10 (extremely).
Headache | -24 hours before race, +24 hours after race, +7 days
  Headache, evaluated through Visual Analogue Scale (VAS) scale. The scoring ranges from 0 (not at all) to 10 (extremely).
Fever | Week -3, -2, -1, -24 hours before race, +24 hours, +7 days after race
  Number of fever episodes in a specified period of time
Respiratory symptoms | Week -3, -2, -1, -24 hours before race, +24 hours, +7 days after race
  Number of days with respiratory symptoms
Sleep quality | Baseline, -24 hours before race, +7 days after race
  Sleep quality, evaluated through 10-point scale. The scoring ranges from 0 (the worst quality) to 10 (best quality).
Adverse events | Baseline, week -3, -2, -1, -24 hours before race, +24 hours, +7 days after race
  Registration of adverse events throughout all study period

CONTACTS AND LOCATIONS:
Overall Officials: Salvador Sarrà, PhD, Principal Investigator — Hospital de Cerdanya
Locations (1):
- Hospital de Cerdanya, Puigcerdà, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cano-Contreras AD, Minero Alfaro IJ, Medina Lopez VM, Amieva Balmori M, Remes Troche JM, Espadaler Mazo J, Perez Lopez N. Efficacy of i3.1 Probiotic on Improvement of Lactose Intolerance Symptoms: A Randomized, Placebo-controlled Clinical Trial. J Clin Gastroenterol. 2022 Feb 1;56(2):141-147. doi: 10.1097/MCG.0000000000001456. PMID 33136781
- [Background] de Oliveira EP, Burini RC, Jeukendrup A. Gastrointestinal complaints during exercise: prevalence, etiology, and nutritional recommendations. Sports Med. 2014 May;44 Suppl 1(Suppl 1):S79-85. doi: 10.1007/s40279-014-0153-2. PMID 24791919
- [Background] Lorenzo-Zuniga V, Llop E, Suarez C, Alvarez B, Abreu L, Espadaler J, Serra J. I.31, a new combination of probiotics, improves irritable bowel syndrome-related quality of life. World J Gastroenterol. 2014 Jul 14;20(26):8709-16. doi: 10.3748/wjg.v20.i26.8709. PMID 25024629